CLINICAL TRIAL: NCT00417651
Title: Transgastric Bacterial Contamination of the Abdomen
Brief Title: Testing for Bacterial Contamination During Gastric Surgeries
Status: Completed | Type: Observational
Sponsor: Jeffrey Hazey (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Hazey, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2006H0078
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Gastric Surgery
Keywords: Bacterial; contamination; gastrotomy; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether creating a gastrotomy (hole in the stomach) during gastric surgery increases a patient's risk of intra-abdominal infection.

We hypothesize that a gastrotomy does not contaminate the abdomen with clinically significant bacterial pathogens.

DETAILED DESCRIPTION:
We propose to investigate the bacterial load and contamination patients experience during laparoscopic roux-en-y gastric bypass while having their gastrotomy for gastrojejunostomy. In all patients who undergo laparoscopic roux-en-y gastric bypass, the stomach must be opened to the peritoneal cavity while placing an anvil for gastrojejunostomy.

Samples of gastric fluid will be collected and sent for analysis in all patients. Samples of peritoneal fluid will be collected prior to and after the creation of the gastrotomy, using intraperitoneal irrigation with approximately 500 cc of normal saline. Bacterial counts and identification will be recorded for each sample.

ELIGIBILITY:
Inclusion Criteria:

* any patient undergoing roux-en-y gastric bypass

Exclusion Criteria:

* lack of consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: observational studies patients morbidly obese.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Quantitative and qualitative measure of the bacterial load and bacterial contamination of the abdomen during laparoscopic roux-en-y gastric bypass surgery while the gastrotomy is open to the abdominal cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Hazey, MD, Principal Investigator — OSU; William S Melvin, MD, Principal Investigator — OSU
Locations (1):
- The Ohio State University Center for Minimally Invasive Surgery, Columbus, Ohio, United States